CLINICAL TRIAL: NCT02004262
Title: A Phase 2B, Randomized, Controlled, Multicenter, Open-Label Study of the Efficacy and Immune Response of GVAX Pancreas Vaccine (With Cyclophosphamide) and CRS 207 Compared to Chemotherapy or to CRS-207 Alone in Adults With Previously-Treated Metastatic Pancreatic Adenocarcinoma
Brief Title: Safety and Efficacy of Combination Listeria/GVAX Pancreas Vaccine in the Pancreatic Cancer Setting
Acronym: ECLIPSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aduro Biotech, Inc. (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-04
Record Dates: First submitted 2013-10-23; First posted 2013-12-09 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: 2nd-line, 3rd-line and Greater Metastatic Pancreatic Cancer
Keywords: cancer; cancer vaccine; Listeria monocytogenes; Listeria-based vaccine; GVAX; cyclophosphamide; Cytoxan; immunotherapy; mesothelin
MeSH Terms: conditions — Neoplasms | interventions — Drug Therapy; Cyclophosphamide

ARMS (6):
- Primary Cohort: Cy/GVAX + CRS-207 (Experimental): * 200 mg per square meter (mg/m^2) cyclophosphamide (Cy) administered by intravenous (IV) infusion on Day 1 of Weeks 1 and 4; GVAX pancreas vaccine (GVAX, 5 × 10e8 cells) administered by intradermal injection on Day 2 of Weeks 1 and 4; CRS-207 (1 × 10e9 colony forming units [CFU]) administered by IV infusion on Day 1 of Weeks 7, 10, 13, 16.
  * The Primary Cohort comprised those subjects who failed at least 1 gemcitabine-based regimen administered for pancreatic cancer in any setting and failed at least 2 prior chemotherapy regimens administered for pancreatic cancer in the metastatic setting.
  Interventions: Biological: GVAX Pancreas Vaccine; Biological: CRS-207; Drug: cyclophosphamide
- Primary Cohort: CRS-207 (Experimental): * CRS-207 (1 × 10e9 CFU) administered by IV infusion on Day 1 of Weeks 1, 4, 7, 10, 13, 16.
  * The Primary Cohort comprised those subjects who failed at least 1 gemcitabine-based regimen administered for pancreatic cancer in any setting and failed at least 2 prior chemotherapy regimens administered for pancreatic cancer in the metastatic setting.
  Interventions: Biological: CRS-207
- Primary Cohort: Chemotherapy (Active Comparator): * Investigator's choice of one of the following: gemcitabine (1000 mg/m^2) administered by IV infusion on Days 1, 8, and 15 of a 28-day cycle; capecitabine (1000 mg/m^2) administered orally twice a day on Days 1 through 14 of a 21-day cycle; fluorouracil with or without leucovorin (2400 mg^m2) administered by IV infusion over 46 hours on Days 1 and 15 of a 28-day cycle; irinotecan (150 mg/m^2) administered by IV infusion on Days 1 and 15 of a 28-day cycle; or erlotinib (100 mg) administered orally once a day for a 21-day cycle.
  * The Primary Cohort comprised those subjects who failed at least 1 gemcitabine-based regimen administered for pancreatic cancer in any setting and failed at least 2 prior chemotherapy regimens administered for pancreatic cancer in the metastatic setting.
  Interventions: Drug: Chemotherapy
- 2nd-line Cohort: Cy/GVAX + CRS-207 (Experimental): * 200 mg/m^2 Cy administered by IV infusion on Day 1 of Weeks 1 and 4; GVAX pancreas vaccine (5 × 10e8 cells) administered by intradermal injection on Day 2 of Weeks 1 and 4; CRS-207 (1 × 10e9 CFU) administered by IV infusion on Day 1 of Weeks 7, 10, 13, 16.
  * The 2nd-line Cohort comprised those subjects who received and failed 1 prior chemotherapy regimen administered for pancreatic cancer in the metastatic setting.
  Interventions: Biological: GVAX Pancreas Vaccine; Biological: CRS-207; Drug: cyclophosphamide
- 2nd-line Cohort: CRS-207 (Experimental): * CRS-207 (1 × 10e9 CFU) administered by IV infusion on Day 1 of Weeks 1, 4, 7, 10, 13, 16.
  * The 2nd-line Cohort comprised those subjects who received and failed 1 prior chemotherapy regimen administered for pancreatic cancer in the metastatic setting.
  Interventions: Biological: CRS-207
- 2nd-line Cohort: Chemotherapy (Active Comparator): * Investigator's choice of one of the following: gemcitabine (1000 mg/m^2) administered by IV infusion on Days 1, 8, and 15 of a 28-day cycle; capecitabine (1000 mg/m^2) administered orally twice a day on Days 1 through 14 of a 21-day cycle; fluorouracil with or without leucovorin (2400 mg^m2) administered by IV infusion over 46 hours on Days 1 and 15 of a 28-day cycle; irinotecan (150 mg/m^2) administered by IV infusion on Days 1 and 15 of a 28-day cycle; or erlotinib (100 mg) administered orally once a day for a 21-day cycle.
  * The 2nd-line Cohort comprised those subjects who received and failed 1 prior chemotherapy regimen administered for pancreatic cancer in the metastatic setting.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Biological: GVAX Pancreas Vaccine
  Other Names: GVAX
  Arms: 2nd-line Cohort: Cy/GVAX + CRS-207; Primary Cohort: Cy/GVAX + CRS-207
Biological: CRS-207
  Arms: 2nd-line Cohort: CRS-207; 2nd-line Cohort: Cy/GVAX + CRS-207; Primary Cohort: CRS-207; Primary Cohort: Cy/GVAX + CRS-207
Drug: Chemotherapy — Investigator's choice of one of the following commercially available products: gemcitabine; capecitabine; fluorouracil with or without leucovorin; irinotecan; or erlotinib.
  Arms: 2nd-line Cohort: Chemotherapy; Primary Cohort: Chemotherapy
Drug: cyclophosphamide
  Other Names: Cytoxan
  Arms: 2nd-line Cohort: Cy/GVAX + CRS-207; Primary Cohort: Cy/GVAX + CRS-207

SUMMARY:
Test the safety, immune response and efficacy of GVAX pancreas vaccine (with cyclophosphamide) and CRS-207 compared to chemotherapy or CRS-207 alone in adults with previously treated metastatic pancreatic adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Have histologically proven malignant adenocarcinoma of the pancreas; measurable disease is not required, mixed histology is not allowed; subjects must have metastatic disease
* 2nd line, 3rd line or greater
* At least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Anticipated life expectancy >12 weeks
* For women and men of childbearing potential, a medically acceptable method of highly effective contraception (oral hormonal contraceptive, condom plus spermicide, or hormone implants) must be used throughout the study period and for 28 days after their final vaccine administration. A barrier method of contraception must be employed by all subjects (male and female), regardless of other methods.
* Have adequate organ function as defined by specified laboratory values

Exclusion Criteria:

* Allergy to both penicillin & sulfa or suspected hypersensitivity to granulocyte-macrophage colony stimulating factor (GM-CSF), dimethyl sulfoxide, fetal bovine serum, trypsin, yeast, glycerol or other component of the therapy options
* Known history or evidence of brain metastases, immunodeficiency disease or immunocompromised state or history of autoimmune disease requiring systemic steroids or other immunosuppressive treatment
* Have any evidence of hepatic cirrhosis or clinical or radiographic ascites
* Have prosthetic heart valves, major implant or device placed in the last 12 months or history of infection with implant/device that cannot be easily removed
* Rapidly progressing disease
* Clinically significant and/or malignant pleural effusion
* Received prior GVAX pancreas vaccine or CRS-207
* Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug, or planned surgery requiring general anesthesia
* Infection with HIV or hepatitis B or C at screening
* Valvular heart disease that requires antibiotic prophylaxis for prevention of endocarditis
* Pregnant or breastfeeding
* Unable to avoid close contact with another individual known to be at high risk of listeriosis (e.g., newborn infant, pregnant woman, HIV-positive individual) during the course of CRS-207 treatment until completion of antibiotic regimen
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (20):
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - University California San Diego Moores Cancer Center, La Jolla, California
  - University of California Mt Zion Comprehensive Cancer Center, San Francisco, California
  - University of California Los Angeles, Santa Monica, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami/Sylvester Cancer Center, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center Morris Cancer Center, Durham, North Carolina
  - Providence Cancer Center, Portland, Oregon
  - University of Pittsburgh Medical Center Cancer Pavillion, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital Princess Margaret Cancer Center, Toronto, Ontario, Canada

REFERENCES:
- [Background] Brockstedt DG, Giedlin MA, Leong ML, Bahjat KS, Gao Y, Luckett W, Liu W, Cook DN, Portnoy DA, Dubensky TW Jr. Listeria-based cancer vaccines that segregate immunogenicity from toxicity. Proc Natl Acad Sci U S A. 2004 Sep 21;101(38):13832-7. doi: 10.1073/pnas.0406035101. Epub 2004 Sep 13. PMID 15365184
- [Background] Le DT, Brockstedt DG, Nir-Paz R, Hampl J, Mathur S, Nemunaitis J, Sterman DH, Hassan R, Lutz E, Moyer B, Giedlin M, Louis JL, Sugar EA, Pons A, Cox AL, Levine J, Murphy AL, Illei P, Dubensky TW Jr, Eiden JE, Jaffee EM, Laheru DA. A live-attenuated Listeria vaccine (ANZ-100) and a live-attenuated Listeria vaccine expressing mesothelin (CRS-207) for advanced cancers: phase I studies of safety and immune induction. Clin Cancer Res. 2012 Feb 1;18(3):858-68. doi: 10.1158/1078-0432.CCR-11-2121. Epub 2011 Dec 6. PMID 22147941
- [Background] Lutz E, Yeo CJ, Lillemoe KD, Biedrzycki B, Kobrin B, Herman J, Sugar E, Piantadosi S, Cameron JL, Solt S, Onners B, Tartakovsky I, Choi M, Sharma R, Illei PB, Hruban RH, Abrams RA, Le D, Jaffee E, Laheru D. A lethally irradiated allogeneic granulocyte-macrophage colony stimulating factor-secreting tumor vaccine for pancreatic adenocarcinoma. A Phase II trial of safety, efficacy, and immune activation. Ann Surg. 2011 Feb;253(2):328-35. doi: 10.1097/SLA.0b013e3181fd271c. PMID 21217520
- [Background] Laheru D, Lutz E, Burke J, Biedrzycki B, Solt S, Onners B, Tartakovsky I, Nemunaitis J, Le D, Sugar E, Hege K, Jaffee E. Allogeneic granulocyte macrophage colony-stimulating factor-secreting tumor immunotherapy alone or in sequence with cyclophosphamide for metastatic pancreatic cancer: a pilot study of safety, feasibility, and immune activation. Clin Cancer Res. 2008 Mar 1;14(5):1455-63. doi: 10.1158/1078-0432.CCR-07-0371. PMID 18316569
- [Background] Le DT, Wang-Gillam A, Picozzi V, Greten TF, Crocenzi T, Springett G, Morse M, Zeh H, Cohen D, Fine RL, Onners B, Uram JN, Laheru DA, Lutz ER, Solt S, Murphy AL, Skoble J, Lemmens E, Grous J, Dubensky T Jr, Brockstedt DG, Jaffee EM. Safety and survival with GVAX pancreas prime and Listeria Monocytogenes-expressing mesothelin (CRS-207) boost vaccines for metastatic pancreatic cancer. J Clin Oncol. 2015 Apr 20;33(12):1325-33. doi: 10.1200/JCO.2014.57.4244. Epub 2015 Jan 12. PMID 25584002
- [Derived] Le DT, Picozzi VJ, Ko AH, Wainberg ZA, Kindler H, Wang-Gillam A, Oberstein P, Morse MA, Zeh HJ 3rd, Weekes C, Reid T, Borazanci E, Crocenzi T, LoConte NK, Musher B, Laheru D, Murphy A, Whiting C, Nair N, Enstrom A, Ferber S, Brockstedt DG, Jaffee EM. Results from a Phase IIb, Randomized, Multicenter Study of GVAX Pancreas and CRS-207 Compared with Chemotherapy in Adults with Previously Treated Metastatic Pancreatic Adenocarcinoma (ECLIPSE Study). Clin Cancer Res. 2019 Sep 15;25(18):5493-5502. doi: 10.1158/1078-0432.CCR-18-2992. Epub 2019 May 24. PMID 31126960
- See also: The Pancreatic Cancer Action Network's Patient & Liaison Services (PALS) program provides patients and families with information and resources at no cost. Visit www.pancan.org, call 877-272-6226 or email pals@pancan.org for information. — http://www.pancan.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with previously treated metastatic pancreatic adenocarcinoma from 21 medical centers in the United States and Canada. The last patient completed the study in August 2016.
Pre-assignment Details: Participants screened over a 21-day period.
Period: Overall Study
Arm/Group | Primary Cohort: Cy/GVAX + CRS-207 | Primary Cohort: CRS-207 | Primary Cohort: Chemotherapy | 2nd-line Cohort: Cy/GVAX + CRS-207 | 2nd-line Cohort: CRS-207 | 2nd-line Cohort: Chemotherapy
Started | 73 | 68 | 72 | 29 | 31 | 30
Treated | 68 | 58 | 43 | 26 | 29 | 11
Completed (No predetermined study completion date or study completion event specified in protocol.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/death, so no subjects "completed" study.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/death, so no subjects "completed" study.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/death, so no subjects "completed" study.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/death, so no subjects "completed" study.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/death, so no subjects "completed" study.) | 0 (Subjects followed until lost to follow-up/consent withdrawn/death, so no subjects "completed" study.)
Not Completed | 73 | 68 | 72 | 29 | 31 | 30
Not completed — Death | 67 | 64 | 66 | 28 | 29 | 22
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 0 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 4 | 3 | 2 | 1 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Baseline analysis provided for all randomized subjects who were administered at least 1 dose of protocol-specified drug (the Full Analysis Set [FAS]).
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Cohort: Cy/GVAX + CRS-207 | Primary Cohort: CRS-207 | Primary Cohort: Chemotherapy | 2nd-line Cohort: Cy/GVAX + CRS-207 | 2nd-line Cohort: CRS-207 | 2nd-line Cohort: Chemotherapy | Total
Number analyzed (Participants) | 68 | 58 | 43 | 26 | 29 | 11 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.96) | 63.2 (8.92) | 64.0 (10.85) | 63.9 (11.83) | 64.1 (9.43) | 66.6 (10.86) | 63.7 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 26 | 15 | 10 | 5 | 116
  Male | 37 | 29 | 17 | 11 | 19 | 6 | 119

OUTCOME MEASURES:

1. Primary Outcome: Primary Cohort: Overall Survival (OS) Censored at 138 Deaths (ITT Set)
Description: OS was estimated using Kaplan-Meier (KM) methods with 95% confidence intervals (CIs), with censoring at the date when 138 deaths were reached in the Primary Cohort in the FAS. Subjects without documentation of death at the time of final analysis were censored as of the date the subject was last known to be alive on/prior to the primary analysis data cut.
Time Frame: Subjects were followed from date of randomization to the date of death by any cause, whichever came first, assessed up to 32 months. Analysis conducted when 138 deaths reached in the Primary Cohort in the FAS.
Population: Analysis based on subjects in the Primary Cohort in the intent-to-treat (ITT) set. The ITT set is the analysis population that included all randomized study subjects.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Primary Cohort: Cy/GVAX + CRS-207 | Primary Cohort: CRS-207 | Primary Cohort: Chemotherapy
Number analyzed (Participants) | 73 | 68 | 72
months | 3.8 [2.9 to 5.3] | 5.4 [4.2 to 6.9] | 4.6 [4.2 to 5.8]

2. Primary Outcome: Primary Cohort: OS (All Data, FAS)
Description: For all treated subjects, OS was calculated using KM methods with 95% CIs. Subjects without documentation of death at the time of the analysis were censored as of the date the subject was last known to be alive on/prior to the final analysis data cut.
Time Frame: Subjects followed for survival from date of randomization until lost to follow-up, withdrawal of consent, or death, whichever came first, assessed up to 32 months.
Population: Analysis based on subjects in the Primary Cohort in the FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Primary Cohort: Cy/GVAX + CRS-207 | Primary Cohort: CRS-207 | Primary Cohort: Chemotherapy
Number analyzed (Participants) | 68 | 58 | 43
months | 4.2 [3.0 to 5.4] | 5.2 [4.2 to 6.3] | 4.7 [3.8 to 6.0]

3. Primary Outcome: 2nd-line Cohort: OS (All Data, FAS)
Description: For all treated subjects, OS was calculated using KM methods with 70% CIs. Subjects without documentation of death at the time of the analysis were censored as of the date the subject was last known to be alive on/prior to the final analysis cut. 70% CIs were selected to provide an 80% probability to rule out differences in median survival less than -2.4 months between the 2nd-line Cohort: Chemotherapy arm and the 2nd-line Cohort: Cy/GVAX + CRS-207 and 2nd-line Cohort: CRS-207 arms, based upon the assumptions made in the statistical analysis plan (SAP).
Time Frame: as for outcome 2
Population: Analysis based on subjects in the 2nd-line Cohort in the FAS.
Measure: Median (70% Confidence Interval); unit: months
Arm/Group | 2nd-line Cohort: Cy/GVAX + CRS-207 | 2nd-line Cohort: CRS-207 | 2nd-line Cohort: Chemotherapy
Number analyzed (Participants) | 26 | 29 | 11
months | 4.6 [3.9 to 6.0] | 4.0 [3.4 to 6.7] | 6.9 [4.2 to 12.3]

4. Secondary Outcome: Number of Participants With Adverse Events in Each Treatment Arm Treatment Regimen
Description: Safety was assessed based upon the number of adverse events (AEs) that occurred in the FAS of each treatment arm, including serious AEs and total AEs. Total AEs included both serious and non-serious AEs.
Time Frame: From the start of the first study drug administration on Day 1, Week 1, through 28 days after the last study drug dose, assessed up to 32 months from the date of randomization.
Population: Analysis conducted for the FAS of each study arm.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Cohort: Cy/GVAX + CRS-207: * 200 mg/m^2 Cy administered by IV infusion on Day 1 of Weeks 1 and 4; GVAX pancreas vaccine (5 × 10e8 cells) administered by intradermal injection on Day 2 of Weeks 1 and 4; CRS-207 (1 × 10e9 CFU) administered by IV infusion on Day 1 of Weeks 7, 10, 13, 16.
  * Participants from both the Primary and 2nd-Line Cohorts receiving at least 1 Cy/GVAX + CRS-207 treatment were combined to form the Pooled Cohort.
- Pooled Cohort: CRS-207: * CRS-207 (1 × 10e9 CFU) administered by IV infusion on Day 1 of Weeks 1, 4, 7, 10, 13, 16.
  * Participants from both the Primary and 2nd-Line Cohorts receiving at least 1 CRS-207 treatment were combined to form the Pooled Cohort.
- Pooled Cohort: Chemotherapy: * Investigator's choice of one of the following: gemcitabine (1000 mg/m^2) administered by IV infusion on Days 1, 8, and 15 of a 28-day cycle; capecitabine (1000 mg/m^2) administered orally twice a day on Days 1 through 14 of a 21-day cycle; fluorouracil with or without leucovorin (2400 mg^m2) administered by IV infusion over 46 hours on Days 1 and 15 of a 28-day cycle; irinotecan (150 mg/m^2) administered by IV infusion on Days 1 and 15 of a 28-day cycle; or erlotinib (100 mg) administered orally once a day for a 21-day cycle.
  * Participants from both the Primary and 2nd-Line Cohorts receiving at least 1 chemotherapy treatment were combined to form the Pooled Cohort.
Arm/Group | Pooled Cohort: Cy/GVAX + CRS-207 | Pooled Cohort: CRS-207 | Pooled Cohort: Chemotherapy
Number analyzed (Participants) | 94 | 87 | 54
Participants
  Serious AEs | 44 | 32 | 15
  Total AEs | 94 | 87 | 52

ADVERSE EVENTS:
Time Frame: From the start of the first study drug administration on Day 1, Week 1, through 28 days after the last study drug dose, assessed up to 32 months from the date of randomization.
Description: Adverse events reported for the FAS study population. Study data were not compiled for other (not including serious) adverse events as an individual category. Therefore, the reported data in the "Other (Not Including Serious) Adverse Events" section includes all adverse events reported in the study and occurring with a 5% or greater frequency, including both serious and non-serious adverse events.
Arm/Group | Pooled Cohort: Cy/GVAX + CRS-207 | Pooled Cohort: CRS-207 | Pooled Cohort: Chemotherapy
All-Cause Mortality (participants affected / at risk) | 88/94 | 82/87 | 51/54
Serious Adverse Events (participants affected / at risk) | 44/94 | 32/87 | 15/54
Other Adverse Events (participants affected / at risk) | 94/94 | 87/87 | 51/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Cohort: Cy/GVAX + CRS-207 (N=94) | Pooled Cohort: CRS-207 (N=87) | Pooled Cohort: Chemotherapy (N=54)
Abdominal Pain (Gastrointestinal disorders) | 4 | 4 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 13 | 5 | 2
Pyrexia (General disorders) | 1 | 1 | 1
Death (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Device dislocation (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 3 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastrointestinal anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Cohort: Cy/GVAX + CRS-207 (N=94) | Pooled Cohort: CRS-207 (N=87) | Pooled Cohort: Chemotherapy (N=54)
Chills (General disorders) | 59 | 81 | 5
Pyrexia (General disorders) | 51 | 58 | 9
Fatigue (General disorders) | 50 | 38 | 26
Vaccination site erythema (General disorders) | 77 | 0 | 0
Vaccination site induration (General disorders) | 53 | 0 | 0
Vaccination site pain (General disorders) | 53 | 0 | 0
Vaccination site oedema (General disorders) | 51 | 0 | 0
Vaccination site pruritus (General disorders) | 49 | 0 | 0
Vaccination site bruising (General disorders) | 25 | 0 | 0
Oedema peripheral (General disorders) | 15 | 6 | 2
Disease progression (General disorders) | 13 | 5 | 2
Pain (General disorders) | 8 | 7 | 2
Asthenia (General disorders) | 5 | 3 | 2
Vaccination site vesicles (General disorders) | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 42 | 44 | 29
Vomiting (Gastrointestinal disorders) | 32 | 32 | 13
Abdominal pain (Gastrointestinal disorders) | 30 | 33 | 12
Constipation (Gastrointestinal disorders) | 25 | 21 | 10
Diarrhoea (Gastrointestinal disorders) | 12 | 18 | 20
Abdominal pain upper (Gastrointestinal disorders) | 8 | 4 | 4
Abdominal distension (Gastrointestinal disorders) | 9 | 4 | 2
Flatulence (Gastrointestinal disorders) | 8 | 5 | 2
Ascites (Gastrointestinal disorders) | 8 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 24 | 16 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 10 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 7 | 3
Dehydration (Metabolism and nutrition disorders) | 8 | 6 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 9 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 6 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 17 | 20 | 1
Blood alkaline phosphatase increased (Investigations) | 18 | 13 | 2
Alanine aminotransferase increased (Investigations) | 12 | 16 | 1
Weight decreased (Investigations) | 10 | 6 | 3
Blood bilirubin increased (Investigations) | 8 | 3 | 2
Blood albumin decreased (Investigations) | 5 | 7 | 0
Lymphocyte count decreased (Investigations) | 7 | 4 | 1
Blood creatinine increased (Investigations) | 6 | 4 | 0
Blood sodium decreased (Investigations) | 5 | 4 | 0
International normalised ratio increased (Investigations) | 5 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 19 | 18 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 10 | 4
Leukocytosis (Blood and lymphatic system disorders) | 5 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3
Hypotension (Vascular disorders) | 18 | 18 | 0
Hypertension (Vascular disorders) | 10 | 13 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 13 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 11 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1
Headache (Nervous system disorders) | 18 | 19 | 2
Dizziness (Nervous system disorders) | 7 | 10 | 3
Neuropathy peripheral (Nervous system disorders) | 3 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 11
Erythema (Skin and subcutaneous tissue disorders) | 8 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Tachycardia (Cardiac disorders) | 13 | 15 | 2
Sinus tachycardia (Cardiac disorders) | 3 | 6 | 1
Insomnia (Psychiatric disorders) | 9 | 5 | 2
Confusional state (Psychiatric disorders) | 5 | 4 | 2
Anxiety (Psychiatric disorders) | 2 | 5 | 3
Urinary tract infection (Infections and infestations) | 3 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 3
Bile duct obstruction (Hepatobiliary disorders) | 5 | 3 | 1

LIMITATIONS AND CAVEATS:
A high number of patients in the chemotherapy arm withdrew from the study before receiving treatment. This high dropout rate may have an impact on interpretation of the study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less